CLINICAL TRIAL: NCT02326753
Title: Gender and Proper Size of Oropharyngeal Airway: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 4-2014-0805
Record Dates: First submitted 2014-12-22; First posted 2014-12-29 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2014-11

CONDITIONS: Adult Patients Undergoing Surgery That Requires General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- No. 7 oral airway (Experimental)
  Interventions: Device: No. 7 oral airway
- No. 8 oral airway (Experimental)
  Interventions: Device: No. 8 oral airway
- No. 9 oral airway (Active Comparator)
  Interventions: Device: No. 9 oral airway

INTERVENTIONS:
Device: No. 7 oral airway — the use of 7 cm sized-oropharyngeal airway (Guedel-type color coded oropharyngeal airway, Hudson RCI, Teleflex Medical, Research Triangle Park, NC)
  Arms: No. 7 oral airway
Device: No. 8 oral airway — the use of 8 cm sized-oropharyngeal airway (Guedel-type color coded oropharyngeal airway, Hudson RCI, Teleflex Medical, Research Triangle Park, NC)
  Arms: No. 8 oral airway
Device: No. 9 oral airway — the use of 9 cm sized-oropharyngeal airway (Guedel-type color coded oropharyngeal airway, Hudson RCI, Teleflex Medical, Research Triangle Park, NC)
  Arms: No. 9 oral airway

SUMMARY:
The purpose of this study is to assess the adequacy of mask ventilation with the different sized-oropharyngeal airway.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing surgery that requires general anesthesia

Exclusion Criteria:

* anticipated difficult intubation
* patients without teeth or with loose teeth
* cervical spine disease
* body mass index over 35 kg/m2
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
the proportion of patients whose oropharyngeal airway is proper | up to 10 minutes after the start of anesthetic induction
  The oropharyngeal airway will be inserted into the patient's mouth. Investigators will check the laryngeal view using fiberoptic bronchoscope and the adequacy of ventilation after the investigator ventilates the patient using the face mask. If both the laryngeal view and ventilation are appropriate, the size of oropharyngeal airway will be considered as the proper size for the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain MedicineSeverance Hospital, Yonsei University Health System, Seoul, Korea, South Korea